CLINICAL TRIAL: NCT06459479
Title: Conversational Artificial Intelligence Simulations to Improve Non-Technical Skills Among Anesthesiology Trainees: A Prospective, Mixed-Methods Study
Brief Title: Conversational AI Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 75964
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Medical Education
Keywords: artificial intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI Group (Experimental): Participant will be using OpenAI's ChatGPT4o's application. For the purposes of this medical error scenario, the CAI will have a standardized prompt to simulate an upset parent whose child recently had surgery in which there was a medical error involving a tooth injury from an intubation. Following a scripted briefing, simulation will be initiated.
  Interventions: Other: Conversational Artificial Intelligence Simulations

INTERVENTIONS:
Other: Conversational Artificial Intelligence Simulations — Use of Conversational Artificial Intelligence Simulations generate medical scenario.

SUMMARY:
This is a prospective, collaborative, mixed-methods study which includes anesthesiology trainees receiving one active intervention - a conversational artificial intelligence (CAI) simulation. The goal is to explore the capability of AI to provide high-fidelity simulations that can ultimately improve how healthcare professionals handle difficult conversations such as disclosing medical errors or mistakes.

ELIGIBILITY:
Inclusion Criteria:

* Hospital providers, including nurses, physician assistants, physicians, physician trainees, and other healthcare workers at Lucile Packard Children's Hospital (LPCH) and affiliated facilities who communicate with patients daily will be included

Exclusion Criteria:

* Participants with reported severe motion sickness
* Nausea
* Seizure disorder
* Currently using chronotropic heart medications, such as β blockers

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate acceptance of Conversational Artificial Intelligence Simulations using Guided Discussion Interview Question Guide | Before simulation
  Guided Discussion Interview Question Guide contains 6 questions focusing 3 areas including Attitudes and Opinions, Perceptions and Summation question. All the questions are open-ended questions.

SECONDARY OUTCOMES:
Evaluation of Conversational Artificial Intelligence Simulations usability via the System Usability Scale (SUS) | Immediately after simulation
  Measured with the System Usability Scale (SUS). The scale has 10 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
Evaluation of Conversational Artificial Intelligence Simulations usability via the User Experience Questionnaire (UEQ-S). | Immediately after simulation
  UEQ-S, includes eight items (four from the pragmatic scales Efficiency, Perspicuity, Dependability, and four from the hedonic scales Stimulation and Novelty). Scores range from -3 (min) to 3 (max)
Evaluation of the reliability of AI quantitative assessment of non-technical performance compared to expert human assessors | immediately after simulation
  The Anaesthetist Non-Technical Skills (ANTS) tool previously published by Fletcher et al. translated in French. The ANTS scoring system uses four categories assessing task management, teamworking, situation awareness and decision-making (1 to 4 points by categories). The minimum score is 4 and the maximum 16

IPD SHARING:
Plan to Share IPD: No